CLINICAL TRIAL: NCT02689141
Title: Prospective, Open-label, Multicentre Phase-II Trial to Evaluate Efficacy and Safety of a Sequential Regimen of Bendamustine Followed by Ofatumumab and Ibrutinib Followed by Ibrutinib and Ofatumumab Maintenance in CLL Patients
Brief Title: Sequential Regimen of Bendamustin-Debulking Followed by Ofatumumab and Ibrutinib in CLL Patients (CLL2-BIO)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: German CLL Study Group (Other)
Collaborators: Gilead Sciences (Industry); Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLL2-BIO; 2014-000590-39 (EudraCT Number)
Record Dates: First submitted 2016-01-29; First posted 2016-02-23 (Estimated); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: chronic lymphocytic leukemia CLL; untreated chronic lymphocytic leukemia; relapsed chronic lymphocytic leukemia; refractory chronic lymphocytic leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, B-Cell | interventions — Bendamustine Hydrochloride; ofatumumab; ibrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bendamustine + Ofatumumab + Ibrutinib (Experimental): Bendamustine: 70mg/m² i.v. Ofatumumab: 1000 mg i.v. Ibrutinib: 420 mg po
  Interventions: Drug: Bendamustine; Drug: Ofatumumab; Drug: Ibrutinib

INTERVENTIONS:
Drug: Bendamustine — Debulking: Cycles 1 - 2, d1 & 2: 70 mg/m2 i.v.
Drug: Ofatumumab — Induction:
  Cycle 1: Day 1 300 mg i.v.; Day 8 1000 mg i.v.; Day 15 1000 mg i.v. Cycle 2-6: Day 1 1000 mg i.v.
  Maintenance: After the induction ofatumumab iv 1000 mg every three months will be continued.
  Cycle 1-8: Day 1 1000 mg i.v.
Drug: Ibrutinib — Induction: Cycle 2-6: d1-28: 420 mg p.o. Maintenance: After the induction ibrutinib p.o. 420 mg daily will be continued. Cycle 1-8: d1-84: 420 mg p.o.

SUMMARY:
A prospective, open-label, multicentre phase-II trial to evaluate the efficacy and safety of a sequential regimen of bendamustine followed by ofatumumab and ibrutinib followed by ibrutinib and ofatumumab maintenance in CLL patients.

DETAILED DESCRIPTION:
In the CLL2-BIO trial an allcomer CLL population with indication for treatment will be included.

Patient will receive 2 cycles of debulking treatment with bendamustin unless contraindications are existing or debulking is not indicated. Afterwards 6 cycles of induction therapy with ofatumumab and ibrutinib will be applied, each with a duration of 28 days. Primary endpoint overall Response rate will be assessed at final restaging.

Patients benefitting from BIO treatment will enter the maintenance phase of the trial. Maintenance treatment will be continued if no unacceptable toxicity occurs until three months after negativity of minimal residual disease (MRD) is achieved in peripheral blood in patients with (clinical) complete response (CR) or (clinical) incomplete complete response (CRi) confirmed by 2 consecutive testings of MRD within 3 months, progression of CLL, start of a subsequent therapy or up to 8 cycles of maintenance (each cycle with a duration of 84 calendar days = 3 months), whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

1. Documented CLL requiring treatment (irrespective if first- or relapse treatment) according to International Working Group on CLL (iwCLL) criteria

   In case of previously treated patients, these must have recovered from acute toxicities and treatment regimen must be stopped within the following time periods before start of the study treatment in the CLL2-BIO trial:
   * chemotherapy within ≥ 28 days
   * antibody treatment within ≥ 14 days
   * kinase inhibitors, Bcl-2-antagonists or immunomodulatory agents within ≥ 3 days
   * corticosteroids may be applied until the start of the BIO-regimen, these have to be reduced to an equivalent of ≤ 20 mg prednisolone during treatment
2. Adequate hematologic function as indicated by a platelet count ≥ 25 x 109/L, a neutrophil count ≥ 1,0 x 109/L and a hemoglobin value ≥ 8.0 g/dL, unless directly attributable to the patient´s CLL (e.g. bone marrow infiltration)
3. Adequate renal function as indicated by a creatinine clearance ≥ 30ml/min calculated according to the modified formula of Cockcroft and Gault or directly measured with 24 hrs urine collection
4. Adequate liver function as indicated by a total bilirubin ≤ 2x, aspartate aminotransferase (AST)/ alanin aminotransferase (ALT) ≤ 2.5x the institutional upper limit of normal (ULN) value, unless directly attributable to the patient's CLL or to Gilbert's Syndrome
5. Negative serological testing for hepatitis B, negative testing for hepatitis-C RNA and negative HIV antibody test within 6 weeks prior to registration
6. Age ≥ 18 years
7. Eastern Cooperative Oncology Group (ECOG) Performance Status 0 to 2, ECOG 3 is only permitted if related to CLL (e.g. due to anemia or severe constitutional symptoms)
8. Life expectancy ≥ 6 months
9. Ability and willingness to provide written informed consent and to adhere to the study visit schedule and other protocol requirements

Exclusion Criteria:

1. Transformation of CLL (i.e. Richter's transformation, pro-lymphocytic leukemia)
2. Known central nervous system (CNS) involvement
3. Patients with confirmed progressive multifocal leukoencephalopathy (PML)
4. Malignancies other than CLL currently requiring systemic therapy
5. Uncontrolled infection requiring systemic treatment
6. Any comorbidity or organ system impairment rated with a cumulative illness rating scale (CIRS) score of 4, excluding the eyes/ears/nose/throat/larynx organ system or any other life- threatening illness, medical condition or organ system dysfunction that - in the investigator´s opinion - could compromise the patients safety or interfere with the absorption or metabolism of the study drugs (e.g, inability to swallow tablets or impaired resorption in the gastrointestinal tract)
7. Use of investigational agents which might interfere with the study drug within 3 days prior to Registration
8. Known hypersensitivity to ofatumumab, ibrutinib or any of the excipients Please note: Patients with a known hypersensitivity to bendamustine are allowed to participate but will not receive a debulking with bendamustine
9. Requirement of treatment with strong CYP3A4-inhibitors/-inducers or anticoagulant with phenprocoumon (marcumar), warfarin, or other vitamin k antagonists
10. History of stroke or intracranial hemorrhage within 6 months prior to registration
11. Pregnant women and nursing mothers (a negative pregnancy test is required for all women of childbearing potential within 7 days before start of treatment and monthly during debulking, induction and maintenance therapy)
12. Fertile men or women of childbearing potential unless:

    * surgically sterile or ≥ 2 years after the onset of menopause, or
    * willing to use two methods of reliable contraception including one highly effective (Pearl Index < 1) and one additional effective (barrier) method during study treatment and for 12 months after end of study treatment.
13. Vaccination with a live vaccine ≤ 28 days prior to registration
14. Legal incapacity
15. Prisoners or subjects who are institutionalized by regulatory or court order
16. Persons who are in dependence to the sponsor or an investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2016-02-04 (Actual); Primary Completion 2017-07-13 (Actual); Study Completion 2020-02-06 (Actual)

PRIMARY OUTCOMES:
Overall response rate (ORR) | 84 days after first dose of last induction cycle
  Proportion of patients responding according to international working Group on chronic lymphocytic leukemia criteria

SECONDARY OUTCOMES:
Safety: Adverse events (AEs) and adverse events of special interest (AESI) | up to 48 months after first dose of study drug
  Type, frequency, and severity of adverse events (AEs) and adverse events of special interest (AESI) and their relationship to study treatment.
minimal residual disease (MRD) | up to 48 months after first dose of study drug
  Rate of MRD responses in peripheral blood measured by immunophenotyping

CONTACTS AND LOCATIONS:
Overall Officials: Paula Cramer, Dr.med., Principal Investigator — German CLL Study Group
Locations (1):
- German CLL Study Group, Cologne, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Langerbeins P, Giza A, Robrecht S, Cramer P, von Tresckow J, Al-Sawaf O, Fink AM, Furstenau M, Kutsch N, Simon F, Goede V, Hoechstetter M, Niemann CU, da Cunha-Bang C, Kater A, Dubois J, Gregor M, Staber PB, Tausch E, Schneider C, Stilgenbauer S, Eichhorst B, Fischer K, Hallek M. Reassessing the chronic lymphocytic leukemia International Prognostic Index in the era of targeted therapies. Blood. 2024 Jun 20;143(25):2588-2598. doi: 10.1182/blood.2023022564. PMID 38620092
- [Derived] Cramer P, Tausch E, von Tresckow J, Giza A, Robrecht S, Schneider C, Furstenau M, Langerbeins P, Al-Sawaf O, Pelzer BW, Fink AM, Fischer K, Wendtner CM, Eichhorst B, Kneba M, Stilgenbauer S, Hallek M. Durable remissions following combined targeted therapy in patients with CLL harboring TP53 deletions and/or mutations. Blood. 2021 Nov 11;138(19):1805-1816. doi: 10.1182/blood.2020010484. PMID 34086865
- [Derived] Cramer P, Tresckow JV, Robrecht S, Bahlo J, Furstenau M, Langerbeins P, Pflug N, Al-Sawaf O, Heinz WJ, Vehling-Kaiser U, Durig J, Tausch E, Hensel M, Sasse S, Fink AM, Fischer K, Kreuzer KA, Bottcher S, Ritgen M, Kneba M, Wendtner CM, Stilgenbauer S, Eichhorst B, Hallek M. Bendamustine, followed by ofatumumab and ibrutinib in chronic lymphocytic leukemia (CLL2-BIO): primary endpoint analysis of a multicenter, open-label phase-II trial. Haematologica. 2021 Feb 1;106(2):543-554. doi: 10.3324/haematol.2019.223693. PMID 32107341